CLINICAL TRIAL: NCT01705704
Title: An Exploratory Evaluation of Interleukin 28B (IL28B) Genotype, Single Nucleotide Polymorphisms (SNP) of rs12356193, Protein and RNA Biomarkers in Serum Samples (Stored, Already Obtained From Completed Studies) From Subjects With HBe-antigen Positive or Negative Chronic Hepatitis B, Who Have Completed Therapy for Hepatitis B With Pegasys ± Lamivudine.
Brief Title: A Retrospective Biomarker Study of Stored Samples Obtained From Patients With Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BV28333
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This retrospective study will evaluate the association of biomarkers and the treatment response of patients with chronic hepatitis B, who have completed therapy with Pegasys (peginterferon alfa-2a) ± lamivudine. For the analysis stored serum samples obtained from patients will be used; no actual patients are involved.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HBe-antigen positive or negative chronic hepatitis B, and no other chronic viral infections who completed therapy for Hepatitis B with Pegasys ± lamivudine
* Inclusion criteria relevant to the clinical studies WV16240, WV16241, and Neptune/WV19432
* Samples from patients treated with either Pegasys or Pegays + lamivudine are included in this analytical study
* Samples will only be analyzed for patients where Investigational Review Board approval has been granted

Exclusion Criteria:

* Exclusion criteria relevant to the clinical studies WV16240, WV16241, and Neptune/WV19432

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stored serum samples obtained from patients with chronic hepatitis B, who have completed therapy with Pegasys +/- lamivudine.
Sampling Method: Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Interleukin-28B (IL-28B) genotype in stored serum samples of patients with chronic hepatitis B, who have completed therapy with Pegasys +/- lamivudine | Samples up to 72 weeks of treatment
Single nucleotide polymorphisms (SNP) of rs12356193 in stored serum samples of patients with chronic hepatitis B, who have completed therapy with Pegasys +/- lamivudine | Samples up to 72 weeks of treatment

SECONDARY OUTCOMES:
IL-28B concentration at baseline and during treatment with Pegasys +/- lamivudine from stored serum samples of patients with chronic hepatitis B | Samples up to 72 weeks of treatment
Protein/RNA biomarker evaluation from stored serum samples of patients with chronic hepatitis B, who have completed therapy with Pegasys +/- lamivudine | Samples up to 72 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Australia (2):
  - Herston, Queensland
  - Fitzroy, Victoria
- Clichy, France
- Hong Kong, Hong Kong
- Italy (4):
  - Bari, Apulia
  - Brescia, Lombardy
  - Cagliari, Sardinia
  - Pisa, Tuscany
- New Zealand (2):
  - Auckland
  - Hamilton
- Russia (3):
  - Saint Petersburg
  - Samara
  - Stavropol
- Singapore, Singapore
- Seoul, South Korea
- Taiwan (3):
  - Kaohsiung City
  - Taipei
  - Taoyuan District
- Thailand (4):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
  - Songkhla

REFERENCES:
- [Derived] van Bommel F, van Bommel A, Krauel A, Wat C, Pavlovic V, Yang L, Deichsel D, Berg T, Bohm S. Serum HBV RNA as a Predictor of Peginterferon Alfa-2a Response in Patients With HBeAg-Positive Chronic Hepatitis B. J Infect Dis. 2018 Aug 24;218(7):1066-1074. doi: 10.1093/infdis/jiy270. PMID 29741634